CLINICAL TRIAL: NCT06346639
Title: Time Course of Adaptive Responses in Humans During a 16-day Hot and Cold Acclimation Program, and Its Effect on Health-related Indicators
Brief Title: Effect of a 16-day Hot and Cold Acclimation on Adaptive Responses and Health-related Indicators
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LithuananianSportsU-17
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Hot Temperature

STUDY DESIGN:
Masking Description: The researchers who will analyze the saliva and venous blood samples will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 16-day hot and cold acclimation (Experimental): Healthy young subjects will participate in a 16-days hot and cold acclimation program. During cold procedure, the participant will be immersed in 14° water bath in semi recumbent position up to the level of the manubrium for 5-min, and during hot procedure, the participant will be immersed in 45° water bath in semi recumbent position up to the level of the manubrium for 5-min.
  Interventions: Other: 16-day hot and cold acclimation

INTERVENTIONS:
Other: 16-day hot and cold acclimation — Acclimation program will consist of 8 brief cold water immersions (CWI; 14°C 5 min) and 8 hot water immersions (HWI; 45°C 5 min). Heat and cold sessions will be performed on separate days (i.e., 1st day hot exposure, 2nd day cold exposure, 3rd day hot exposure, etc.).

SUMMARY:
There are no previous studies of the effects of a combination of whole-body immersions in hot and cold baths on adaptive responses and health-related markers. Thus, the primary aim of this project is to determine whether interventions consisting of whole body immersion in hot and cold baths over 16 days develop heat and/or cold adaptation by remodeling thermoregulatory, metabolic, cardiovascular and physiological responses, and the secondary aim is to determine if current cold-hot acclimation has any effects on physical and mental health-related markers.

ELIGIBILITY:
Inclusion Criteria:

* young, healthy, non-obese males and females;
* nonsmoker;
* no needle phobia;
* not taking medication and/or dietary supplements that may affect experimental variables.

Exclusion Criteria:

* neurological, cardiovascular, metabolic, and/or inflammatory diseases, or conditions that could be worsened by exposure to acute thermal stimuli and that could affect experimental variables;
* involvement in temperature manipulation program for ≥ 3 months;
* attendance at any excessive formal physical exercise or sports program.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2029-04-04 (Estimated); Study Completion 2029-04-04 (Estimated)

PRIMARY OUTCOMES:
Change in body mass and body composition (kg) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Body mass and composition (in kg) will be evaluated using Tanita Body Composition Analyzer (Japan).
Change in skinfold thickness (mm) | Before acclimation (1st day), 2 days and 2 weeks after the end of acclimation (44 th and 51st day)
  Skinfolds thickness (in mm) will be measured using a skinfold caliper (Saehan, Korea) at 10 sites and the mean subcutaneous fat thickness will be calculated.
Change in body mass index (kg/m^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The body mass index (in kg/m^2) will be defined as the body mass divided by the square of the body height.
Change in body surface area (m^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The participant's body surface area (BSA) (in m^2) will be estimated using the following equations: BSA = 128.1 ×weight^0.44 × height^0.60 for males and BSA = 147.4 ×weight^0.47 × height^0.55 for females.
Change in substrate oxidation | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Oxygen consumption (VO2) and carbon dioxide (VCO2) output will be measured using Cortex METALYZR® 3B, Leipcig, Germany), and the respiratory quotient (RQ = VCO2 / VO2) will be computed to determine substrate utilisation. The RQ values for fat is assumed as 0.7, for protein is assumed as 0.8 and for carbohydrate isassumed as 1.0.
Change in substrate oxidation (g/day) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Carbohydrate and fat oxidation (in g/day) will be measured using Cortex METALYZR® 3B, Leipcig, Germany).
Change in ventilation (l/min) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Ventilation (in l/min) will be measured using Cortex METALYZR® 3B, Leipcig, Germany).
Change in breathing frequency (t/min) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Breathing frequency (in t/min) will be measured using Cortex METALYZR® 3B, Leipcig, Germany).
Change in resting energy expenditure (kcal/day) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The resting energy expenditure (REE; in kcal/day) will be computed using the following equation: REE = [3.941 × (VO2) + 1.106 × (VCO2)] × 1440
Change in metabolic heat production (W) | during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days)
  The metabolic heat production (MHP; in W) will be computed using the equation: MHP = (281.65 + 80.65 × RQ) × VO2.
Change in heart rate (bpm) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Heart rate (in bpm) will be recorded using a heart rate sensor with a chest strap (Polar, Finland) or Physioflow hemodynamic monitor (France).
Change in blood pressure (mmHg) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Systolic and diastolic blood pressure (in mmHg) will be measured using PROVIEW 10 Compact Patient Monitor (Germany).
Change in mean arterial pressure (mmHg) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The mean arterial pressure (MAP; in mmHg) will be estimated using the formula: MAP = DP + 1/3(SP - DP) or MAP = DP + 1/3(SP - DP), where SP is systolic bood pressure and DP is diastolic blood pressure.
Change in heart rate variability (ms) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  R-R intervals (in ms) in supine resting will be recorded using a Polar heart ratesensor (Finland) and simultaneously transferred to Polar Pro Trainer 5 software (Finland)
Change in heart rate variability (time domain) (ms) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Heart rate variability data will be analyzed using Kubios heart rate variability analysis software (Finland). In the time domain that reflects general heart rate variability (HRV), the standard deviation of normal-to-normal intervals (SDNN; estimate of overall HRV) and the root mean square of successive differences (RMSSD; estimate of short-term components of HRV will be assessed (in ms).
Change in heart rate variability (time domain) (Ln) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Heart rate variability data will be analyzed using Kubios heart rate variability analysis software (Finland). In the time domain that reflects general heart rate variability (HRV), the standard deviation of normal-to-normal intervals (SDNN; estimate of overall HRV) and the root mean square of successive differences (RMSSD; estimate of short-term components of HRV) will be assessed and logarithmically transformed (Ln) to correct the skewness of distribution.
Change in heart rate variability (frequency domain) (ms^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Heart rate variability data will be analyzed using Kubios heart rate variability analysis software (Finland). In the frequency domain that measures the more specific contribution of the autonomic nervous system branch, low-frequency (LF; estimates sympathetic and parasympathetic activity) and high-frequency (HF; estimates parasympathetic activity) powers in absolute units (in m^2) will be assessed.
Change in heart rate variability (frequency domain) (Ln) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  In the frequency domain that measures the more specific contribution of the autonomic nervous system branch, low-frequency (LF; estimates sympathetic and parasympathetic activity) and high-frequency (HF; estimates parasympathetic activity) powers will be assessed and logarithmically transformed (Ln) to correct the skewness of distribution.
Change in stroke volume (ml) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Stroke volume (in ml) will be recorded using Physioflow hemodynamic monitor (France).
Change in stroke volume index (ml/m^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Stroke volume index (in ml/m^2) will be recorded using Physioflow hemodynamic monitor (France).
Change in cardiac output index (l/min//m^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Cardiac output (in l/min/m^2) will be recorded using Physioflow hemodynamic monitor (France).
Change in cardiac output index (l/min) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Cardiac output (in l/min) will be recorded using Physioflow hemodynamic monitor (France).
Change in contractility index | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Contractility index will be recorded using Physioflow hemodynamic monitor (France).
Change in ventricular ejection time (ms) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Ventricular ejection time (in ms) will be recorded using Physioflow hemodynamic monitor (France).
Change in ventricular ejection fraction (percent) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Ejection fraction (in percent) will be recorded using Physioflow hemodynamic monitor (France).
Change in end diastolic volume (ml) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  End diastolic volume (in ml) will be recorded using Physioflow hemodynamic monitor (France).
Change in systemic vascular resistance (dyn.s/cm5.m^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Systemic vascular resistance (in dyn.s/cm5.m^2) will be recorded using Physioflow hemodynamic monitor (France).
Change in cardiac work index (kg.m/m^2) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Cardiac work index (in kg.m/m^2) will be recorded using Physioflow hemodynamic monitor (France).
Change in early diastolic filling ratio (percent) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Early diastolic filling ratio (in percent) will be recorded using Physioflow hemodynamic monitor (France).
Change in testosterone concentration (µg/dl) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The saliva samples will be collected to measure testosterone level (in µg/dl) using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).
Change in female sex hormones concentration (pg/mL) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The venous 17beta-estradiol and progesterone (in pg/mL), follicle stimulating hormone and luteinizing hormone will be measured using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).
Change in salivary cortisol concentration (µg/dl) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The saliva samples will be collected to measure cortisol level (in µg/dl) using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria)..
Change in cytokines concentrations (pg/ml) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The venous tumor necrosis factor alpha, interleukin-6 and IL-1 beta (in pg/ml) will be measured using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).
Change in complete blood count (10^9/L) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Complete blood count with 5 different white blood count components (absolute neutrophils, lymphocytes, monocytes, eosinophils, basophils) analysis (in 10^9/L) will be performed using an automated Mythic 60 hematology analyzer (Switzerland).
Change in complete blood count (percent) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Complete blood count with 5 different white blood count components (absolute neutrophils, lymphocytes, monocytes, eosinophils, basophils) analysis (in percent) will be performed using an automated Mythic 60 hematology analyzer (Switzerland).
Change in lipid profile (mmol/l) | Before acclimation (1st day),during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Blood samples will be collected to measure lipid profile (in mmol/l) (total cholesterol, high density and low density cholesterol, triglycerides) using a CardioChek PA analyzer (USA).
Change in catecholamines concentration (ng/ml) | Before acclimation (1st day),during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  The venous adrenaline and noradrenaline concentrations (in ng/ ml) will be measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).
Change in insulin concentration (μIU/ml) | Before acclimation (1st day), 2nd day and 2 weeks after the end of acclimation (44th and 51st days)
  The venous insulin concentrations (in μIU/ml) will be measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria)
Change in glucose tolerance (mmol/l) | Before acclimation (1st day), 2nd day and 2 weeks after the end of acclimation (44th and 51st days)
  The glucose concentration (in mmol/l) will be measured using a On-call GK dual meter (Acon Laboratories, USA).
Change in anxiety and depression (points) | Before acclimation (1st day), 2nd day and 2 weeks after the end of acclimation (44th and 51st days)
  The level of anxiety and depression (in points) will be defined using Hospital Anxiety and Depression scale. Scale scores range from 0 to 21, with higher scores indicating more severe symptoms.
Change in plasma metabolites of the kynurenine pathway (μm) | Before acclimation (1st day), during baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  An ultra-performance liquid chromatography-tandem mass spectrometry system (UPLC-MS/MS) will be used to measure venous plasma levels of tryptophan, kynurenine, kynurenic acid, 3-hydroxy-kynurenine, quinolinic acid, nicotinamide and picolinic acid (in μm). The UPLC-MS/MS system uses a Xevo TQ-XS triple quadrupole mass spectrometer (Waters) with a Z-spray electrospray interface, and the system operates in electrospray positive multiple reaction monitoring mode.
Change in body temperature (°C) | During baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days), and 2 weeks after the end of acclimation (51st day)
  Rectal temperature (in °C) will be measured using a thermocouple (Rectal Probe, Ellab, Denmark) inserted to a depth of 12 cm past the anal sphincter, skin temperature (in °C) will be measured with thermistors (Skin/Surface Probe, DM852, Ellab) at four sites: supraclavicular, back, thigh, and forearm, and right lateral gastrocnemius muscle temperature (in °C) will be measured using a needle microprobe (MKA; Ellab).
Change in physiological strain index | During baseline provocative heat test (8th or 15th day), during acclimation (from 22 to 37th days), during repeated provocative heat test (41st or 42nd days)
  A physiological strain index (PSI) will be used to indicate heat strain. PSI = 5 x (Tret - Tre0) x (39.5 - Tre0)^-1+ 5 x (HRt - HR0) x (180 - HR0)^-1, where rectal temperature (Tre) t and heart rate (HR) t are simultaneous measurements taken at the end of the heat exposure and Tre0 and HR0 are the initial measurements.
Change in cold strain index | During baseline provocative cold test (8th or 15th day), during acclimation (from 22 to 37th days), during repeated provocative cold test (41st or 42nd days)
  A cold strain index (CSI) will be used to indicate cold strain. CSI = 6.67 x (Tre t - Tre 0) x (35 - Tre 0)^-1 + 3.33 x (Tsk t - Tsk 0) x (20 - Tsk 0)^-1, where rectal temperature (Tre) 0 and skin temperature (Tsk) 0 are initial measurements and Tre t and Tsk t are simultaneous measurements taken at the end of the cold exposure.
Change in root mean square (RMS) amplitude (mV) | During baseline provocative cold test (8th or 15th day), during acclimation (from 22 to 37th days), during repeated provocative cold test (41st or 42nd day)
  Root mean square (RMS) amplitude (in mV) of pectoralis major muscle indicating shivering intensity will be measured using a surface EMG (Biometrics, UK).
Change in pain sensations | During baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st or 42nd day)
  The pain sensation will be evaluated using numeric pain scale ranging from 0 (no pain) to 10 (worst possible pain).
Change in thermal sensations (points) | During baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st or 42nd day)
  The thermal sensation will be evaluated using 9-point scale. The rating of thermal sensation range from 1 (very cold) to 9 (very hot), with 5 being neutral.
Change in shivering/sweating (points) | During baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st or 42nd day)
  The shivering/sweating rate will be evaluated using 7-point scale. The rating of shivering/sweating range from 1 (heavily sweating) to 7 (vigorously shivering), with 4 being neutral.
Change in thermal comfort (points) | During baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st or 42nd day)
  The thermal comfort will be evaluated using 4-point scale. The rating of thermal comfort range from 0 (neutral) to 3 (very uncomfortable).

SECONDARY OUTCOMES:
Height (m) | Before acclimation (1st day)
  Height (in m) will be measured using a Harpenden anthropometer set (Holtain Ltd, UK)
Change in physical activity (in h) | 3 days before first assessment, during 16-day acclimation period and during 2 week post-acclimation period.
  MotionWatch 8 actigraph will estimate the time spent in sedentary, light, moderate, or vigorous activity
Change in sleep (in h) | 3 days before first assessment, during 16-day acclimation period and during 2 week post-acclimation period.
  Sleep statistics (in h) including total hours of sleep and the time spent in different sleep stages will be assessed with MotionWatch 8 actigraph.
Change in oxygen saturation (percent) | During baseline provocative tests (8th and 15th day), during acclimation (from 22 to 37th days), during repeated provocative tests (41st and 42nd days)
  Oxygen saturation (in percent) will be measured using Proview 10 Compact Patient Monitor (Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Jarutienė, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No